CLINICAL TRIAL: NCT06749223
Title: AQT90 FLEX D-dimer Clinical Sensitivity and Specificity
Status: Recruiting | Type: Observational
Sponsor: Radiometer Medical ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: DC-078241
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-12

CONDITIONS: VTE (Venous Thromboembolism)
Keywords: D-dimer
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: D-dimer test — Blood sample collection for D-dimer testing

SUMMARY:
The goal of this study is evaluate the clinical performance of the AQT90 FLEX D-dimer Test as an aid in the diagnosis of Venous Thromboembolism.

DETAILED DESCRIPTION:
The objective is to evaluate the clinical performance of the AQT90 FLEX D-dimer Test as an aid in the diagnosis of VTE in patients presenting with low or moderate pretest probability (PTP), by determining the clinical sensitivity, specificity, negative predictive value (NPV), positive predictive value (PPV), positive likelihood ratio (LR+) and negative likelihood ratio (LR-) of the assay.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age and older
* Subject, who presents with signs and symptoms of VTE and had low or moderate pre-test probability of DVT or PE assessed by Well's score
* Subject must be able to understand information given, and be willing and able to voluntarily give their consent to participate in this study

Exclusion Criteria:

* Subject, who is pregnant
* Subject, who has received fibrinolytic therapy within the previous seven days
* Subject, who has received treatment with anticoagulants (unfractionated heparin, LMWH, VKA (vitamin K-antagonists), DOACs (direct oral anticoagulants) within the previous seven days
* Subject, who has had trauma or surgery within the previous four weeks
* Subject with malignancy
* Subject with disseminated intravascular coagulation (DIC)
* Subject, who has an invalid written informed consent or has withdrawn consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients presenting with signs and symptoms of VTE and getting clinical evaluation of the pretest probability of VTE scored as low or moderate corresponding to a Well's score between 0-2 for DVT and between 0-6 for PE.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity | From enrollment to blood sample collection; ~1 hour
  Clinical performance (clinical sensitivity, clinical specificity, Negative Predictive Values (NPV), Positive Predictive Values (PPV), Positive Likelihood Ratio (LR+), Negative Likelihood Ratio (LR-) and 95 % confidence intervals) for the AQT90 FLEX D-dimer assay against the hospital diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Viborg Regional Hospital, Viborg, Denmark

IPD SHARING:
Plan to Share IPD: No